CLINICAL TRIAL: NCT06774313
Title: A Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single Ascending Doses of ABBV-142 in Healthy Adult Subjects and Single Doses of ABBV-142 in Healthy Adult Asian Subjects
Brief Title: A Study to Assess the Adverse Events and How Subcutaneous (SC) Injections and Intravenous (IV) Infusions of ABBV-142 Move Through the Body of Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M25-265
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-142

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part 1: Group 1 (Experimental): Participants will receive ABBV-142 Dose A or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 1: Group 2 (Experimental): Participants will receive ABBV-142 Dose B or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 1: Group 3 (Experimental): Participants will receive ABBV-142 Dose C or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 1: Group 4 (Experimental): Participants will receive ABBV-142 Dose D or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 1: Group 5 (Optional) (Experimental): Participants will receive ABBV-142 Dose TBD or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 2: Group 6 (Experimental): Participants will receive ABBV-142 Dose B or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 2: Group 7 (Experimental): Participants will receive ABBV-142 Dose C or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 3: Group 8 (Experimental): Han Chinese participants will receive ABBV-142, dose to be determined, or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo
- Part 3: Group 9 (Experimental): Japanese participants will receive ABBV-142, dose to be determined, or Placebo on Day 1.
  Interventions: Drug: ABBV-142; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-142 — Intravenous (IV) Infusion
  Arms: Part 1: Group 1; Part 1: Group 2; Part 1: Group 3; Part 1: Group 4; Part 1: Group 5 (Optional); Part 3: Group 8; Part 3: Group 9
Drug: ABBV-142 — Subcutaneous (SC) Injection
  Arms: Part 2: Group 6; Part 2: Group 7
Drug: Placebo — IV Infusion
  Arms: Part 1: Group 1; Part 1: Group 2; Part 1: Group 3; Part 1: Group 4; Part 1: Group 5 (Optional); Part 3: Group 8; Part 3: Group 9
Drug: Placebo — SC Injection
  Arms: Part 2: Group 6; Part 2: Group 7

SUMMARY:
This study is designed to assess the pharmacokinetic properties, safety, tolerability, and immunogenicity of ABBV-142 and determine whether predicted efficacious exposures can be safely achieved in humans.

ELIGIBILITY:
Inclusion Criteria:

All Parts:

• Volunteers in general good health.

Part 3, ONLY:

HAN CHINESE Participants:

* Participant must be first- or second-generation Han Chinese of full Chinese parentage (both parents of Han Chinese descent), residing outside of China. Participants must be in general good health.
* First-generation participants will have been born in China to two parents and four grandparents, who were also born in China, and are of full Chinese descent.
* Second-generation participants born outside of China must have two parents and four grandparents born in China and are of full Chinese descent.

OR

JAPANESE Participants:

* Participant must be first- or second-generation Japanese parentage (both parents of Japanese descent), residing outside of Japan. Participants must be in general good health.
* First-generation participants will have been born in Japan to two parents and four grandparents born in Japan and are of full Japanese descent.
* Second-generation participants born outside of Japan must have two parents and four grandparents born in Japan and are of full Japanese descent.

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Use of tobacco or nicotine-containing products within 180 days prior to the first dose of study drug.
* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Day 120
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Observed Serum Concentration (Cmax) of ABBV-142 | Up to Day 120
  Cmax of ABBV-142 will be assessed.
Time to Cmax (Tmax) of ABBV-142 | Up to Day 120
  Tmax of ABBV-142 will be assessed.
Area Under the Serum Concentration-time Curve (AUC) of ABBV-142 from Time 0 to the Time of Last Measurable Concentration (AUCt) | Up to Day 120
  AUCt of ABBV-142 will be determined.
AUC of ABBV-142 from Time 0 to Infinity (AUCinf) | Up to Day 120
  AUCinf of ABBV-142 will be assessed.
Terminal Phase Elimination Rate Constant (β) of ABBV-142 | Up to Day 120
  Terminal phase elimination rate constant (β) of ABBV-142 will be assessed.
Terminal Phase Elimination Half-life (t1/2) of ABBV-142 | Up to Day 120
  Terminal phase elimination half-life (t1/2) of ABBV-142 will be assessed.
Dose Normalized Cmax of ABBV-142 | Up to Day 120
  Dose normalized Cmax of ABBV-142 will be assessed.
Dose Normalized AUC of ABBV-142 | Up to Day 120
  Dose normalized AUC of ABBV-142 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 271899, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-265